CLINICAL TRIAL: NCT00451360
Title: Evaluation of the CHOndromodulating Effect of DIAcerein in Osteoarthritis of the Hip. ECHODIAH.
Brief Title: Chondromodulating Effect of Diacerein in Osteoarthritis of the Hip
Acronym: ECHODIAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires NEGMA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEC / CHO 90040N; AFSSAPS number: 930289; CCPPRB number: 469
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2007-03

CONDITIONS: Hip Osteoarthritis
Keywords: Diacerein; Hip osteoarthritis; Structure-modifying effect / Chondromodulating effect; Double blind study
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: diacerein

SUMMARY:
We carried out a 3 years, randomized, double-blind, placebo-controlled, multicenter clinical trial in patients with hip osteoarthritis in order to:

* evaluate the ability of diacerein, an interleukin-1β inhibitor, to slow the progressive decrease in joint space width observed in patients with hip osteoarthritis
* to investigate the potential structure-modifying effect of diacerein in patients with hip osteoarthritis

This study compare also after ten years the percentage of patients in each treatment group who require a hip replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* Outpatients fulfilling the American College of Rheumatology criteria for the diagnosis of hip osteoarthritis.
* Lequesne algofunctional index of at list 3 points.
* Radiographic criterion for inclusion: joint space width (JSW) between 1 mm and 3 mm. If the JSW exceeded 3 mm, it had to be at least 0.5 mm thinner than JSW of the contra lateral hip, measured at its narrowest point.

Exclusion Criteria:

* Intraarticular injection or arthroscopy of the hip during the three months prior to inclusion in the study.
* Any systemic or intraarticular corticosteroid as well as other potential symptom-modifying drugs for osteoarthritis were not allowed during the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1993-03; Study Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Joint space measurement

SECONDARY OUTCOMES:
Requirement of hip replacement surgery after ten years
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: DOUGADOS Maxime, Principal Investigator — Scientific committee; Michel LEQUESNE, Principal Investigator — Scientific committee; Bernard MAZIERE, Principal Investigator — Scientific committee; Eric VIGNON, Principal Investigator — Scientific committee; Laurent BERDAH, Principal Investigator — Scientific committee; Minh NGUYEN, Principal Investigator
Locations (25):
- France (25):
  - Hôpital Nord, Amiens
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne
  - CHU cote de Nacre, Caen
  - Hôpital Mondor, Créteil
  - Hôpital Général, Dijon
  - CHU, Grenoble
  - Hôpital Roger Salengro, Lille
  - CHRU Dupuytren, Limoges
  - Hôpital de la Timone, Marseille
  - Hôpital Lapeyronie, Montpellier
  - Hôpital de l'Archet, Nice
  - Hôpital Cochin, clinique de rhumatologie, Paris
  - Paris
  - Hôpital Cochin, Paris
  - Hôpital Leopold Bellan, Paris
  - CH Lyon Sud, Pierre-Bénite
  - CHU Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie, Poitiers
  - CHR, Rennes
  - Hôpitam de Bois Guillaume, Rouen
  - Hôpital de Hautepierre, Strasbourg
  - CHU de Rangueil, Toulouse
  - CHU Trousseau, Tours
  - CHU de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Dougados M, Nguyen M, Berdah L, Mazieres B, Vignon E, Lequesne M; ECHODIAH Investigators Study Group. Evaluation of the structure-modifying effects of diacerein in hip osteoarthritis: ECHODIAH, a three-year, placebo-controlled trial. Evaluation of the Chondromodulating Effect of Diacerein in OA of the Hip. Arthritis Rheum. 2001 Nov;44(11):2539-47. doi: 10.1002/1529-0131(200111)44:113.0.co;2-t. PMID 11710710